CLINICAL TRIAL: NCT05725577
Title: Rheum@Home: Rheumatoid Arthritis Care in the 21th Century
Brief Title: Rheum@Home: RA Remote Patient Monitoring
Acronym: R@H
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: App company failed to produce a working application
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: University of Twente (Other); Reade Rheumatology Research Institute (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Harald E. Vonkeman, Principle Investigator, Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R@H
Record Dates: First submitted 2022-12-13; First posted 2023-02-13 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care via the telemedicine system (Other): Intervention
  Interventions: Other: care via the telemedicine system
- Standard care (Other): Control
  Interventions: Other: Routine care

INTERVENTIONS:
Other: care via the telemedicine system — Care via the telemedicine system
  Arms: Care via the telemedicine system
Other: Routine care — Routine care
  Arms: Standard care

SUMMARY:
The goal of this pragmatic multicentre clinical trial is to investigate whether telemonitoring with Rheum@Home leads to less outpatient visits, while maintaining tight disease control and high patient-experienced quality of care in patients with rheumatoid arthritis.

Participants will be asked to

* complete questionaires every 4 weeks
* perform a walking test every 4 weeks
* routine lab
* routine disease activity measurement by a qualified assessor

Researchers will compare care via the telemedicine system (intervention) or standard care (control) to see if there are differences in the number of rheumatology outpatient visits and patient reported quality of care after 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients;
* signed, written informed consent;
* 18 -75 years of age;
* clinical diagnosis of RA;
* ≥ 6 months stable low disease activity or remission, according to the treating rheumatologist;
* able to read and understand simple Dutch language instructions;
* ownership or access to a smartphone, tablet or computer and having internet access;
* able to conduct a teleconsultation on a smartphone, tablet or computer.

Exclusion Criteria:

* severe comorbidity or other factors necessitating continuation of regular outpatient visits, according to the treating rheumatologist

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Number of rheumatology outpatient visits with rheumatologists and nurses | 12 month period
  Number of rheumatology outpatient visits with rheumatologists and nurses
Patient-reported quality of care | 12 month period
  measured with visual analogue scale (VAS) scores (0-10; higher score indicates higher quality) in seven relevant domains: patients' satisfaction with health care, patients' experiences contacting their health-care providers, the extent to which health care meets patients' expectations, healthcare workers' timeliness of response to questions and symptoms, health-care workers' fulfilment of agreements, health-care workers attentiveness to acute situations, and hospital accessibility in case of symptoms. A mean score of 8 out of 10 or higher was predefined as perceived high quality

SECONDARY OUTCOMES:
Number of rheumatology teleconsultations (email, telephone, video) | 12 month period
  Number of rheumatology teleconsultations (email, telephone, video)
DAS28 | 12 month period
  Disease Activity Score
PROMs: disease activity score (RAPID3) | 12 month period
  PROMs: disease activity score (RAPID3)
PROMs: Patient acceptable symptom state (PASS) | 12 month period
  PROMs: Patient acceptable symptom state (PASS)
PROMs: participation (WPAI) | 12 month period
  PROMs: participation (WPAI)
PROMs: pain (NRS) | 12 month period
  PROMs: pain (NRS)
PROMs: fatigue (NRS) | 12 month period
  PROMs: fatigue (NRS)
PROMs: physical function (HAQ-DI) | 12 month period
  PROMs: physical function (HAQ-DI)
PROMs: health related quality of life (EQ5D) | 12 month period
  PROMs: health related quality of life (EQ5D)
PROMs: health related quality of life (SF36) | 12 month period
  PROMs: health related quality of life (SF36)
Physical performance: 50 meter walking test | 12 month period
  Physical performance: 50 meter walking test
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 month period
  (S)AE's assessed by CTCAE v4.0
Cost-effectiveness: healthcare utilization questionnaire | 12 month period
  Cost-effectiveness: healthcare utilization questionnaire
Patient experience: System usability scale (SUS) | 12 month period
  Patient experience: System usability scale (SUS)
Patient experience: Perceived efficacy in patient-physician interactions (PEPPI-5) | 12 month period
  Patient experience: Perceived efficacy in patient-physician interactions (PEPPI-5)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Vonkeman, MD, Principal Investigator — University of Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol
Time Frame: After publication
Access Criteria: Upon reasonable request to p.m.tenklooster@utwente.nl